CLINICAL TRIAL: NCT06763731
Title: Optimizing the Ocular Surface With Systane COMPLETE in Patients With Dry Eye Planning for Cataract Surgery
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Collaborators: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 202311109MIPD
Record Dates: First submitted 2024-12-12; First posted 2025-01-08 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-10

CONDITIONS: Ophthalmology
Keywords: Dry eye; Cataract surgery
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Intervention Model Description: Prospective, single-arm study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental group (Experimental): Prospective, single-arm study
  Interventions: Drug: Systane COMPLETE

INTERVENTIONS:
Drug: Systane COMPLETE — Preop dry eye management using Systane COMPLETE can help to optimize the ocular surface.
  Other Names: Experimental group

SUMMARY:
Regular use of Systane COMPLETE in dry eye subjects before cataract surgery may optimize the ocular surface.

DETAILED DESCRIPTION:
STUDY OBJECTIVE：To evaluate the impact of predicted residual astigmatism in mixed dry eye patients regularly using Systane COMPLETE before cataract surgery.

Hypothesis：Regular use of Systane COMPLETE in mixed dry eye subjects before cataract surgery may lead to more accurate astigmatism predictions.

Objectives：To evaluate the Impact of predicted residual astigmatism in mixed dry eye patients regularly using Systane COMPLETE before cataract surgery.

Inclusion Criteria The subjects aged 20-85 years, with normal cognitive function and capable of answering related questionnaires who require phacoemulsification and intraocular lens implantation under topical anaesthesia, are the eligible candidates.

Exclusion Criteria Unable to answer the questions in the dry eye survey. Ocular trauma or ocular surgery in the planned surgical eye, active ocular infection, and obvious abnormalities in ocular surface or eyelid margins other than MGD cause decreased visual acuity other than cataracts.

Dry eye signs: Corneal Fluorescein Staining CFS (+) to exclude any corneal abnormalities or epithelial defect.

Systemic drug use, including tetracycline derivatives, antihistamines, and isotretinoin.

Using dry eye medication at screening stage.

Research Process V1 Screening (1-2 month before surgery) The subjects' demographic information will be collected. The pre-op assessments will be performed, and Informed Consent will be explained and endorsed during this visit.

Systane COMPLETE MD1 bottle will be prescribed to all subjects who signed the ICF, with a dosing frequency of 1-2 drops q.i.d OU for 1-2 month.

The LENSTAR 900 device (Haag-Streit Swiss) will be used to measure the biometry of the anterior cornea's keratometry at each visit. The measurement will be taken through five consecutive scans with only a few seconds of interval between each scan. The mean keratometry of these five scans will be used.

Anterior corneal surface maps from Pentacam (OCULUS, Germany) will be used to identify patients with keratoconus or corneal irregularities at each visits.

V2 Pre-operative (7 days before surgery) All participants will receive refractive examinations and take dry eye assessments.

Repeat the same biometry measurement as the first visit. The final choice of the IOL for surgery is based on biometry measurements and Barrett Toric calculation.

One eye per subject will be analysed.

V3 Surgery day The participants will receive phacoemulsification and intraocular lens implantation. The participants with any intra-operative complication will be excluded from the study.

To ensure compliance with the medication, it is required that the subjects return the used Systane COMPLETE bottle and medication diary at V3.

ELIGIBILITY:
Inclusion Criteria:

The subjects aged 20-85 years, with normal cognitive function and capable of answering related questionnaires who require phacoemulsification and intraocular lens implantation under topical anaesthesia, are the eligible candidates.

Exclusion Criteria:

1. Unable to answer the questions in the dry eye survey.
2. Ocular trauma or ocular surgery in the planned surgical eye, active ocular infection, and obvious abnormalities in ocular surface or eyelid margins other than MGD cause decreased visual acuity other than cataracts.
3. Dry eye signs: Corneal Fluorescein Staining CFS (+) to exclude any corneal abnormalities or epithelial defect
4. Systemic drug use, including tetracycline derivatives, antihistamines, and isotretinoin.
5. Using dry eye medication at screening stage

Ages: 20 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2024-05-02 (Actual); Primary Completion 2026-01-15 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
OSDI Dry Eye Questionnaire | 1-2 months
  The Ocular Surface Disease Index (OSDI) questionnaire is a tool designed to evaluate dry eye symptoms, focusing on three aspects: self-reported eye discomfort, visual function impairment, and environmental triggers. The questionnaire contains 12 items, each rated on a scale from 0 to 4, with a total score ranging from 0 to 100. Higher scores indicate more severe dry eye symptoms. The OSDI questionnaire has high reliability and validity, aiding healthcare professionals in quickly assessing the severity of dry eye, making it suitable for clinical diagnosis and treatment evaluation.
Preoperative Assessments for Cataract Surgery at NTUH: Vision Measurement | 1-2 months
  Vision measurement is a core component of the preoperative baseline assessment, providing information on the patient's uncorrected and corrected visual acuity. This data helps determine the necessity of surgery and establish postoperative vision expectations.
Preoperative Assessments for Cataract Surgery at NTUH: Biometry | 1-2 months
  Biometry is an essential part of the preoperative evaluation, providing critical measurements that guide the selection of the appropriate intraocular lens. This assessment ensures precise surgical planning and contributes to achieving optimal visual outcomes postoperatively.
Preoperative Assessments for Cataract Surgery at NTUH: Pentacam(Corneal topography maps) | 1-2 months
  Pentacam is a vital component of the preoperative assessment, offering detailed corneal mapping that aids in evaluating corneal structure and detecting any abnormalities. This information supports surgical planning and enhances the accuracy of intraocular lens selection, contributing to improved postoperative visual outcomes.
K5 (Non-Invasive Tear Break-Up Time (NITBUT)) | 1-2 months
  K5 (Non-Invasive Tear Break-Up Time (NITBUT)) is used to evaluate tear film stability, a key diagnostic indicator for dry eye. It is crucial for enhancing postoperative visual quality.

CONTACTS AND LOCATIONS:
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan, Taiwan